CLINICAL TRIAL: NCT01985932
Title: A Prospective Study Evaluating Non-Endorectal Coil Functional MRI Identification of Intraprostatic Tumor During Radiation Treatment Planning
Brief Title: Functional MRI Use in Prostate Radiation Treatment Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 07812
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Functional MRI (Other): Subjects in this arm receive functional MRI during radiation therapy treatment planning.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI

SUMMARY:
This study is being done to evaluate the use of MRI during radiation treatment planning to identify areas of tumor within the prostate to aid in future treatment planning and targeting of prostate cancer. This study will be conducted at the University of Pennsylvania Health System. The study is projected to run for 18 months. Subjects will be male 18 or older with a prostate cancer diagnosis and treatment plansat the Department of Radiation Oncology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Male
* Biopsy proven prostate cancer without evidence of metastatic disease
* Planned definitive external beam RT with daily ERB and implanted Visicoil fiducial markers.
* Prior fMRI-ec documenting an IPL 25 mm2 in axial bidimensional diameter product, concordant with intraprostatic tumor location as documented on transrectal ultrasoundbiopsy
* Subject capable of giving informed consent for standard external beam RT and for the study.
* No current contraindication that would prevent MRI or gadolinium contrast.

Exclusion Criteria:

* Metastatic disease
* Lack of fMRI-ec documeneting an IPL 25 mm2 in axial bidimensional product, concordant with intraprostatic tumor location as documented on transrectal untrasound biopsy
* Neoadjuvant androgen deprivation therapy greater than 10 weeks, defined from date of LHRH analog injection to date of fMRI-sim
* Contraindication that would prevent MRI or gadolinium contrast
* GFR 30 mL/min/1.73m2 per Crockoft-Gault formula.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtiland Deville, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Functional MRI: Subjects in this arm receive functional MRI during radiation therapy treatment planning.
  MRI
Period: Overall Study
Arm/Group | Functional MRI
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Functional MRI
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.36 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Functional MRI
Number analyzed (Participants) | 15
Participants | 0

ADVERSE EVENTS:
Arm/Group | Functional MRI
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes